CLINICAL TRIAL: NCT04008303
Title: Outcomes of Following Surgical Decompression for the Treatment of Migraine
Brief Title: Outcomes of Migraine Surgery
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled since this study open. The Primary research member (medical school student) is no longer available to do this study
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Brian Drolet, Assistant Professor Department of Plastic Surgery, Vanderbilt University Medical Center
Other Study IDs: 190993
Record Dates: First submitted 2019-06-11; First posted 2019-07-05 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with migraines: Patients seen in clinic and assessed with Migraine Headache Diagnostic Criteria to ensure diagnosis.
  Patients track the characteristics of migraine headaches for one month before surgery.
  After this month, patients receive surgery in the operating room for migraine.
  After surgery, patients track the characteristics of migraine headaches for 3 months.
  Patients will then be asked to track the characteristics migraine headaches again at 1 year and 2 years and 5 years after surgery. For these time periods, patients only have to keep track of the characteristics for 1 month intervals.
  Interventions: Procedure: Migraine surgery

INTERVENTIONS:
Procedure: Migraine surgery — Surgical decompression of neuromuscular structures causing migraine headaches.

SUMMARY:
Migraines are very common and affect over 35 million Americans a year. Migraines can be painful and affect daily life. The cause of migraine is multifactorial and not completely understood. Treatment usually includes different classes of medications, life style changes, physical therapy, acupuncture, nerve stimulators and avoiding common triggers (like bright lights, certain foods, or loud sounds).

For some patients, Botox injected into the muscles of the forehead and neck can significantly reduce pain. Unfortunately, this does not provide long-term relief as the effect of Botox lasts for 3 months. Since year 2000 surgery to treat a selected population of migraine patients has been gaining popularity and showing promising results. The surgery reduces the pressure on the peripheral nerves that are believed to cause migraine headaches by resecting the surrounding tissue (bone, fascia, muscle, and arteries). This surgery provides a more long-term and permanent relief.

The purpose of this study is to follow the effectiveness and outcomes of migraine surgery.

DETAILED DESCRIPTION:
Migraines are very common and affect over 35 million Americans a year. Migraines can be painful and affect daily life. The cause of migraine is multifactorial and not completely understood. Treatment usually includes different classes of medications, life style changes, physical therapy, acupuncture, nerve stimulators and avoiding common triggers (like bright lights, certain foods, or loud sounds).

For some patients, Botox injected into the muscles of the forehead and neck can significantly reduce pain. Unfortunately, this does not provide long-term relief as the effect of Botox lasts for 3 months. Since year 2000 surgery to treat a selected population of migraine patients has been gaining popularity and showing promising results. The surgery reduces the pressure on the peripheral nerves that are believed to cause migraine headaches by resecting the surrounding tissue (bone, fascia, muscle, and arteries). This surgery provides a more long-term and permanent relief.

The purpose of this study is to follow the effectiveness and outcomes of migraine surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Cleared by neurology and headache specialists for surgery
* Patient cleared by neurology for not having medication overuse headaches
* Patient able to localize a consistent trigger site where the migraines start
* Patient has been suffering from migraine for more than 2 years
* Botox injections or nerve blocks have worked for migraine relief in the past
* Patients formally diagnosed with migraine headaches by a neurologist
* Migraines impact quality of life per MIDAS survey
* No history of Mania, Bipolar disorder, Major Dispersive disorder, or suicidal ideation

Exclusion Criteria:

* High dose opioid medication use
* Does not meet criteria for migraine diagnosis
* History of prior surgery for migraines

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with migraine headaches that meet above inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change in International Classification of Headache Disorders Diagnostic criteria: Frequency | 1 month intervals at 1 month, 1 year, 2 years, and 5 years post-operative
  Frequency
  * Number of migraine headaches per day
  * Number of migraine headaches per week
Change in International Classification of Headache Disorders Diagnostic criteria: Duration | 1 month intervals at 1 month, 1 year, 2 years, and 5 years post-operative
  Duration
  -How long the migraine headaches last in minutes
Change in International Classification of Headache Disorders Diagnostic criteria: Location | 1 month intervals at 1 month, 1 year, 2 years, and 5 years post-operative
  Location
  * Area of head that hurts with migraines.
  * Options include front, side, top, and back.
Change in International Classification of Headache Disorders Diagnostic criteria: Quality | 1 month intervals at 1 month, 1 year, 2 years, and 5 years post-operative
  Quality
  * Description of the migraine pain.
  * Options include sharp, stabbing, dull, pulsating, and burning.
Change in International Classification of Headache Disorders Diagnostic criteria: Severity | 1 month intervals at 1 month, 1 year, 2 years, and 5 years post-operative
  Severity
  - Migraine headache severity graded on a 0-10 scale, with 10 being the most severe.
Change in International Classification of Headache Disorders Diagnostic criteria: Laterality | 1 month intervals at 1 month, 1 year, 2 years, and 5 years post-operative
  Laterality
  * Side of the head that is impacted with migraine headaches
  * Options include right, left, or both.
Change in International Classification of Headache Disorders Diagnostic criteria: Associated Symptoms | 1 month intervals at 1 month, 1 year, 2 years, and 5 years post-operative
  Associated symptoms
  * Question to record associated symptoms that occur with migraine headaches
  * Options include nausea, vomiting, photophobia, photophobia, and aura symptoms
Change in International Classification of Headache Disorders Diagnostic criteria: Exacerbating factors | 1 month intervals at 1 month, 1 year, 2 years, and 5 years post-operative
  Exacerbating factors
  * Open ended question to record anything that makes the migraine headaches worse.
  * Examples include medications, environmental triggers (light, noise, etc), and lifestyle (stress, exercise, etc)
Change in International Classification of Headache Disorders Diagnostic criteria: Relieving factors | 1 month intervals at 1 month, 1 year, 2 years, and 5 years post-operative
  Relieving factors
  * Open ended question to record anything that makes the migraine headaches better.
  * Examples include medications, avoidance of environmental triggers (light, noise, etc), and lifestyle changes (stress avoidance, exercise, etc)

CONTACTS AND LOCATIONS:
Overall Officials: Salam Kassis, MD, Study Director — Vanderbilt University Medical Center

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared

REFERENCES:
- [Background] Negro A, Rocchietti-March M, Fiorillo M, Martelletti P. Chronic migraine: current concepts and ongoing treatments. Eur Rev Med Pharmacol Sci. 2011 Dec;15(12):1401-20. PMID 22288302
- [Background] Janis JE, Barker JC, Javadi C, Ducic I, Hagan R, Guyuron B. A review of current evidence in the surgical treatment of migraine headaches. Plast Reconstr Surg. 2014 Oct;134(4 Suppl 2):131S-141S. doi: 10.1097/PRS.0000000000000661. PMID 25254996
- [Background] Stewart WF, Simon D, Shechter A, Lipton RB. Population variation in migraine prevalence: a meta-analysis. J Clin Epidemiol. 1995 Feb;48(2):269-80. doi: 10.1016/0895-4356(94)00128-d. PMID 7869073
- [Background] Leonardi M, Steiner TJ, Scher AT, Lipton RB. The global burden of migraine: measuring disability in headache disorders with WHO's Classification of Functioning, Disability and Health (ICF). J Headache Pain. 2005 Dec;6(6):429-40. doi: 10.1007/s10194-005-0252-4. Epub 2005 Dec 15. PMID 16388337
- [Background] Guyuron B, Kriegler JS, Davis J, Amini SB. Five-year outcome of surgical treatment of migraine headaches. Plast Reconstr Surg. 2011 Feb;127(2):603-608. doi: 10.1097/PRS.0b013e3181fed456. PMID 20966820
- [Background] Gfrerer L, Guyuron B. Surgical treatment of migraine headaches. Acta Neurol Belg. 2017 Mar;117(1):27-32. doi: 10.1007/s13760-016-0731-1. Epub 2016 Dec 24. PMID 28013487
- [Background] Guyuron B, Reed D, Kriegler JS, Davis J, Pashmini N, Amini S. A placebo-controlled surgical trial of the treatment of migraine headaches. Plast Reconstr Surg. 2009 Aug;124(2):461-468. doi: 10.1097/PRS.0b013e3181adcf6a. PMID 19644260
- [Result] Guyuron B, Varghai A, Michelow BJ, Thomas T, Davis J. Corrugator supercilii muscle resection and migraine headaches. Plast Reconstr Surg. 2000 Aug;106(2):429-34; discussion 435-7. doi: 10.1097/00006534-200008000-00030. PMID 10946944
- [Result] Lee M, Monson MA, Liu MT, Reed D, Guyuron B. Positive botulinum toxin type a response is a prognosticator for migraine surgery success. Plast Reconstr Surg. 2013 Apr;131(4):751-757. doi: 10.1097/PRS.0b013e3182818b7f. PMID 23542247
- [Result] Guyuron B, Kriegler JS, Davis J, Amini SB. Comprehensive surgical treatment of migraine headaches. Plast Reconstr Surg. 2005 Jan;115(1):1-9. PMID 15622223